CLINICAL TRIAL: NCT02141633
Title: Airway and Pulmonary Vascular Endothelial Function in Healthy Smokers: Effect of Inhaled Glucocorticosteroid Treatment
Acronym: smoker3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Adam Wanner, Research Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 20120896; NCT02026375 (obsolete NCT alias)
Record Dates: First submitted 2014-03-25; First posted 2014-05-19 (Estimated); Results first posted 2016-12-16 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-10

CONDITIONS: Smoking
Keywords: smokers; airway blood flow; fluticasone; echocardiogram
MeSH Terms: conditions — Smoking | interventions — Albuterol; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- smokers (Experimental): participants with smoking history ( > 10 pack/year) will be enrolled and perform airway blood flow and echocardiogram before and 15 minutes after albuterol inhalation
  Interventions: Procedure: echocardiogram plus albuterol; Procedure: airway blood flow plus albuterol; Drug: Fluticasone propionate; Drug: placebo
- non-smokers (Experimental): healthy life-time non smokers will be enrolled and perform airway blood flow and echocardiogram before and 15 minutes after albuterol inhalation
  Interventions: Procedure: echocardiogram plus albuterol; Procedure: airway blood flow plus albuterol

INTERVENTIONS:
Procedure: echocardiogram plus albuterol — participants will performed echocardiogram before and 15 minutes after inhaled albuterol
Procedure: airway blood flow plus albuterol — participants will performed echocardiogram before and 15 minutes after inhaled albuterol
  Other Names: Qaw
Drug: Fluticasone propionate — participant will be received a 4-week course of inhaled fluticasone (220 μg fluticasone twice a day administered as a MDI using a spacer)
  Arms: smokers
Drug: placebo — participant will be received a 4-week course of identically appearing placebo (2 puffs twice a day via spacer).
  Arms: smokers

SUMMARY:
The purposes of the present proposal are to 1) compare inhaled albuterol-induced changes in airway blood flow (Qaw), and in CO and Ppas in healthy current smokers and lifetime non-smokers as an index of endothelial function in the airway and pulmonary circulations, 2) compare the results between smokers and non-smokers, and 3) determine the effect of a 4-week treatment with an ICS on albuterol responsiveness of Qaw and the echocardiographic parameters. With this protocol the Investigators will test the hypotheses that a) there is a correlation between airway and pulmonary vascular endothelial function within the current smoker and non-smoker groups, and b) ICS treatment improves airway and pulmonary vascular endothelial function in the current smoker group.

DETAILED DESCRIPTION:
With this protocol the Investigators will test the hypotheses that a) there is a correlation between airway and pulmonary vascular endothelial function within the current smoker and non-smoker groups, and b) ICS treatment improves airway and pulmonary vascular endothelial function in the current smoker group.

Fifteen healthy current smokers with a >10 pack-year history of smoking and 15 healthy never-smokers will be enrolled. Males and females between 25 and 75 years of age will be recruited There will be 1-4 visits to the laboratory (one for non-smokers, 4 for smokers). All subjects will have the first visit. Current smokers will have 3 additional visits. Current smokers will be asked not to smoke before coming to the laboratory on the 3 study days. All subjects will be instructed to abstain from ingesting alcoholic beverages, coffee or caffeinated drinks for at least 12 hours the night before each study day. The subjects will also be instructed not to use PDE5 inhibitors for 24 hours before coming to the laboratory. On each study day, the protocol will start at the same time (in the morning).

ELIGIBILITY:
Inclusion Criteria:

* Fifteen healthy current smokers with a >10 pack-year history of smoking and 15 healthy never-smokers will be enrolled. Males and females between 25 and 75 years of age will be recruited.

Exclusion Criteria:

* Women of childbearing potential who do not use accepted birth control measures; pregnant and breast feeding women
* Cardiovascular disease and/or use of cardiovascular medications
* Subjects with known beta-adrenergic agonist intolerance
* A physician diagnosis of chronic airway disease (asthma, COPD, bronchiectasis, cystic fibrosis)
* Acute respiratory infection within four weeks prior to the study
* Use of any airway medication
* Abnormal pulmonary function

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-04; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wanner, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami School of Medicine, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Smokers: participants will performed airway blood flow and echocardiogram before and 15 minutes after inhalation of albuterol.
  echocardiogram: participants will performed echocardiogram before and 15 minutes after inhaled albuterol
  airway blood flow: participants will performed echocardiogram before and 15 minutes after inhaled albuterol
- Non-smokers: participants will performed airway blood flow and echocardiogram before and 15 minutes after inhalation of albuterol
  echocardiogram: participants will performed echocardiogram before and 15 minutes after inhaled albuterol
  airway blood flow: participants will performed echocardiogram before and 15 minutes after inhaled albuterol
Period: Overall Study
Arm/Group | Smokers | Non-smokers
Started | 16 | 15
Completed | 15 | 15
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Smokers; Non-smokers: echocardiogram: participants will performed echocardiogram before and 15 minutes after inhaled albuterol
  airway blood flow: participants will performed echocardiogram before and 15 minutes after inhaled albuterol
- Total: Total of all reporting groups
Arm/Group | Smokers | Non-smokers | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (2.0) | 44.7 (2.0) | 46.2 (2.0)
Gender [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Airway Blood Flow
Description: compare inhaled albuterol-induced changes in airway blood flow (ΔQaw) in healthy current smokers and lifetime non-smokers as an index of endothelial function in the airway circulation and to compare the results between smokers and non-smokers
Time Frame: before and 15 minutes after albuterol inhalation
Measure: Mean (Standard Error); unit: ΔQaw (ul/min/ml)
Arm/Group | Smokers | Non-smokers
Number analyzed (Participants) | 15 | 15
ΔQaw (ul/min/ml) | 2.13 (2.52) | 13.05 (1.22)

2. Secondary Outcome: Echocardiogram
Description: to compare inhaled albuterol-induced changes in echocardiogram measuring mean pulmonary artery pressure (MPAP)in healthy current smokers and lifetime non-smokers as an index of endothelial function in the pulmonary circulation and to compare the results between smokers and non-smokers
Time Frame: MPAP before and 15 minutes after albuterol inhalation in smokers vs non-smokers
Measure: Mean (Standard Error); unit: ΔMPAP (mmHg)
Arm/Group | Smokers | Non-smokers
Number analyzed (Participants) | 15 | 15
ΔMPAP (mmHg) | -7.70 (1.37) | -9.04 (0.74)

ADVERSE EVENTS:
Time Frame: 2 years and 10 month
Groups:
- Smokers; Non-smokers: No AE or SAE had occurred
Arm/Group | Smokers | Non-smokers
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No